CLINICAL TRIAL: NCT00601341
Title: Effects of Lumbosacral Joint Mobilization/Manipulation on Lower Extremity Muscle Neuromuscular Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Anticipated that results would not be conclusive
Sponsor: University of Virginia (Other)
Collaborators: National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other)
Responsible Party: Christopher Ingersoll, PhD, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11730
Record Dates: First submitted 2008-01-14; First posted 2008-01-28 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Knee Pain; Hip Pain; Ankle Pain; Lumbopelvic Pain
Keywords: arthralgia; joint pain; knee injuries; knee joint; low back pain
MeSH Terms: conditions — Arthralgia; Knee Injuries; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): lumbosacral joint manipulation
  Interventions: Other: lumbosacral joint manipulation
- 2 (Experimental): lumbar passive range of motion
  Interventions: Other: lumbar passive range of motion
- 3 (Other): lie on exam table for 3 minutes
  Interventions: Other: No active intervention

INTERVENTIONS:
Other: lumbosacral joint manipulation — lumbosacral joint manipulation
  Arms: 1
Other: lumbar passive range of motion — lumbar passive range of motion
  Arms: 2
Other: No active intervention — Lie on exam table for 3 minutes
  Arms: 3

SUMMARY:
The purpose of this study is to gain a better understanding of the effects of lumbopelvic manual therapy on lower extremity biomechanics and arthrogenic muscle response. As a result of this study, we also hope that physical therapists, athletic trainers, and other physical medicine rehabilitation providers will gain a better understanding of lower extremity injuries and have the scientific evidence to provide patients with techniques which would allow for efficient return to activities of daily living without restrictions and possibly prevent future injuries and minimize risk of osteoarthritis.

The objectives of this study are to:

* Determine the amount and duration of arthrogenic muscle response of quadriceps muscles following lumbopelvic joint manipulation.
* Determine the effects of lumbopelvic joint manipulation on temporospatial parameters of gait such cadence, step length, velocity and mean peak lower extremity joint moments.
* Determine if a correlation exists between patellofemoral joint pain and lumbopelvic joint dysfunction.
* Determine the amount of change in clinical outcome measure scores following lumbopelvic joint manipulation.

DETAILED DESCRIPTION:
It is well known that musculoskeletal dysfunction at one joint is not limited to the joint itself and can be related to dysfunction at joints proximal or distal in the kinetic chain. Recent research has focused on the relationship of altered lower extremity kinematics and common musculoskeletal pathologies.

Pain is often associated with musculoskeletal pathologies and is one of the strongest stimuli affecting functional activities in a negative manner. Following injury or chronic dysfunction, inhibitory neurons decrease the ability of musculature to fully recruit excitatory motor neurons. This can lead to aberrant movement patterns and different activation of muscles. Muscle inhibition has been attributed as a possible source of altered motor activation patterns. Pain can be a result or cause of musculoskeletal dysfunction and does not necessarily precede inhibition, but can have a contributing effect. The presence of muscle inhibition is considered a limiting factor in the rehabilitation of musculoskeletal pathologies. If muscle inhibition is properly addressed, individuals and athletes alike, should be able to more appropriately meet the demands of the activities with a decreased risk of future injury.

One technique used to determine presence of muscle inhibition is to measure the ability of the muscle to produce a maximal voluntary isometric contraction and compare values with the ability of the contralateral muscle. Since the contralateral limb may also experience muscle inhibition,it is difficult to obtain an accurate measurement of the amount of muscle inhibition occurring in the ipsilateral limb. A suggested solution is utilize the burst-superimposition technique which provides the muscle with a supramaximal stimulus to recruit any remaining muscle fibers which have not been stimulated.

Treatment of muscle inhibition is multifaceted. Utilization of manual therapy techniques such as joint manipulation or mobilization directed at the lumbopelvic region have been shown to be successful in disinhibiting lower extremity muscles. Previous studies have demonstrated sacroiliac joint manipulation disinhibited the quadriceps muscle in individuals with anterior knee pain. One of the limitations was these studies only observed an immediate decrease of quadriceps inhibition and the duration of the treatment effect was unknown. Effects of disinhibition of other lower extremity muscles and duration of disinhibition have not been determined at this time. It is also unknown what effects manual therapy treatments directed at the lumbopelvic region have on functional activities such as walking, squatting, or ascending/descending stairs. By examining these effects, we will be attempting to provide scientific evidence to validate common clinical practices in rehabilitative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Physician referral to physical therapy for treatment of insidious onset of lumbopelvic or lower extremity musculoskeletal dysfunction or individuals with chronic lumbopelvic or lower extremity musculoskeletal dysfunction not wishing to seek physical therapy services.

  * Unilateral or Bilateral hip pain or dysfunction
  * Unilateral or Bilateral knee pain or dysfunction with two of the following symptoms:
* Pain reproduced with patella compression, squatting, prolonged sitting, going up or down stairs, or isometric quadriceps contraction.

  * Unilateral or Bilateral ankle pain or dysfunction
  * Lumbopelvic pain or dysfunction
* Control subjects who volunteer in response to advertisements will have healthy, pain free, back, hips, knees, and ankles.

Exclusion Criteria:

* Participants who are outside of age range (to ensure bony maturity while reducing the prevalence of age related degenerative changes and hypomobility.)
* Participants with knee pain which does not fit inclusion criteria.

  * Ligamentous insufficiency, meniscus damage, patellar tendonitis, history of subluxation/dislocation
* Participants with signs indicating nerve root compression (contraindication for lumbopelvic joint manipulation)

  * Pain extending below knee
  * Positive Straight Leg Raise
  * Decreased lower extremity manual muscle test (Below 4/5), decreased sensation, hyporeflexia
* Participants demonstrating upper motor neuron signs (contraindication to lumbopelvic manipulation)

  * Hyperreflexia
  * Pathological reflexes
* Participants who have had lower extremity or spine surgery
* Participants who are unable to run for 5 minutes.
* Participants with ankylosing spondylitis (contraindication for lumbopelvic manipulation)
* Participants with spinal hypermobility or spondylolisthesis. (contraindication for lumbopelvic manipulation)
* Participants with spinal cord disease or cauda equina. (contraindication for lumbopelvic manipulation)
* Participants with osteoporosis. (contraindication for lumbopelvic joint manipulation)
* Participants with rheumatoid arthritis. (contraindication to lumbopelvic joint manipulation.)
* Participants who may be currently pregnant. (contraindication for electrical stimulation and lumbopelvic joint manipulation.)
* Participants with traumatic spine or lower extremity injury within past 6 months
* Participants who are currently participating or have participated in a lower extremity musculoskeletal rehabilitation program within the past 6 months.
* Participants who have had previous adverse reactions to electrical stimulation (i.e. electrode burns.)
* Participants who have a demand-type cardiac pacemaker (contraindication for electrical stimulation)
* Participants with diagnosis of cancer (current cancer is a contraindication for electrical stimulation and relative contraindication for lumbopelvic joint manipulation)
* Participants who are unable to give consent or are unable to understand procedures of experiment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Neuromuscular response (central activation ratio), characteristics of gait (stride length, step length, etc.), joint moments | All study visits up to day 21

SECONDARY OUTCOMES:
Characteristics of gait (stride length, step length, etc.) | All study visits up to day 21
Orthopedic special tests and questionnaires | Concluding at day 21

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ingersoll, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States